CLINICAL TRIAL: NCT00650624
Title: A Dose-Ranging Study Of Valdecoxib 5 Mg, 10 Mg, And 20 Mg QD Versus Placebo In Patients With OA Of The Knee
Brief Title: A Dose-Ranging Study Of Valdecoxib 5 Mg, 10 Mg, And 20 Mg Once Daily Versus Placebo In Patients With Osteoarthritis Of The Knee (Japan)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VALAJP-8274-156; A3471090
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Osteoarthritis, Knee
Keywords: knee osteoarthritis; Japan
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — valdecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 3 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: valdecoxib — valdecoxib 5 mg tablet by mouth once daily in the morning for 6 weeks
  Arms: Arm 1
Drug: valdecoxib — valdecoxib 10 mg tablet by mouth once daily in the morning for 6 weeks
  Arms: Arm 2
Drug: valdecoxib — valdecoxib 20 mg tablet by mouth once daily in the morning for 6 weeks
  Arms: Arm 3
Drug: placebo — placebo tablet by mouth once daily in the morning for 6 weeks
  Arms: Arm 4

SUMMARY:
To determine the therapeutic dose range of valdecoxib by comparing the efficacy of three dosing regimens (5 mg, 10 mg and 20 mg once daily) with placebo for relief of the signs and symptoms of osteoarthritis of the knee. To assess safety and tolerability of multiple doses of valdecoxib in patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with symptomatic OA of the knee by the American College of Rheumatology (ACR) criteria and a Functional Capacity Classification (FCC) of I - III at Screening Visit and were walking
* At the Baseline visit, eligible patients were to have Patient's Assessment of Arthritis Pain VAS ≥ 40 mm and Patient's & Physician's Global Assessment of Arthritis of "Poor" or "Very Poor"

Exclusion Criteria:

* Patients unable to walk generally

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2003-06; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities) OA Pain Index | screening (Day -14), baseline (week 0), and at weeks 2, 4, and 6 (final visit)

SECONDARY OUTCOMES:
patients' and physicians' and 'categorical' global assessment of arthritis | screening (Day -14), baseline (week 0), and at weeks 2, 4, and 6
WOMAC OA stiffness index | screening (Day -14), baseline (week 0), and at weeks 2, 4, and 6
WOMAC OA physical function index | screening (Day -14), baseline (week 0), and at weeks 2, 4, and 6
WOMAC OA composite index | screening (Day -14), baseline (week 0), and at weeks 2, 4, and 6
WOMAC OA pain index, stiffness index, physical function index, and composite index | screening (Day -14), baseline (week 0), and at weeks 2, 4, and 6
Incidence of and time to withdrawal due to lack of efficacy | weeks 2, 4, and 6
patient's assessment of arthritis pain (Visual Analog Scale, VAS) | screening (Day -14), baseline (week 0), and at weeks 2, 4, and 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- Japan (22):
  - Pfizer Investigational Site, Funabashi, Chiba
  - Pfizer Investigational Site, Sakura, Chiba
  - Pfizer Investigational Site, Chikushi-gun, Fukuoka
  - Pfizer Investigational Site, Iizuka, Fukuoka
  - Pfizer Investigational Site, Kurume, Fukuoka
  - Pfizer Investigational Site, Yame, Fukuoka
  - Pfizer Investigational Site, Chitose, Hokkaido
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Kamakura, Kanagawa
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Isahaya, Nagasaki
  - Pfizer Investigational Site, Hirakata, Osaka
  - Pfizer Investigational Site, Kanzaki-gun, Saga-ken
  - Pfizer Investigational Site, Karatsu, Saga-ken
  - Pfizer Investigational Site, Ogi-gun, Saga-ken
  - Pfizer Investigational Site, Itabashi-ku, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-Ku, Tokyo
  - Pfizer Investigational Site, Taito-ku, Tokyo
  - Pfizer Investigational Site, Yoyogi Shibuya-ku, Tokyo
  - Pfizer Investigational Site, Saga
  - Pfizer Investigational Site, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=VALAJP-8274-156&StudyName=A%20Dose-Ranging%20Study%20of%20Valdecoxib%205%20mg%2C%2010%20mg%2C%20and%2020%20mg%20Once%20Daily%20versus%20Placebo%20in%20Patients%20with%20Osteoarthritis%20of%20th